CLINICAL TRIAL: NCT05730660
Title: Effectiveness of a 3-months Dietary Supplementation Based on Quercetin Phytosome®) for the Treatment of Chronic Fatigue Symptoms
Brief Title: Quercetin Phytosome® Chronic Fatigue Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0912/01072022
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2023-02

CONDITIONS: Chronic Fatigue Symptoms; Sleep; Physical Performance; Body Composition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Dietary Supplement: Quercetin group
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo group

INTERVENTIONS:
Dietary Supplement: Quercetin group — 2 capsules a day of Quercetin Fitosoma® of 250 mg each
  Arms: Intervention group
Dietary Supplement: Placebo group — 2 tablets per day, white film-coated having the same appearance as Quercetin Fitosoma ® tablets.
  Arms: Placebo group

SUMMARY:
The purpose of this study is to evaluate whether a 3-month period of quercetin supplementation (500 mg of Quercetin Phytosome®) is useful in the treatment of chronic fatigue, as assessed by the Fatigue Impact Scale (FIS-40). Secondary end points are sleep assessment through Pittsburgh Sleep Quality Index (PSQI) and muscle performance assessment through the Short Physical Performance Battery (SPPB) and body composition assessment using DXA.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* Chronic fatigue symptoms recorded using a self-reported fatigue score assessed using the validated Fatigue Impact Scale (FIS- 40) that comprised chronic tiredness impacts related to physical, cognitive and psychosocial functions.

Exclusion Criteria:

* Patients with any active medical condition that explains chronic fatigue (untreated hypothyroidism, sleep apnea, narcolepsy, drug side effects, and iron deficiency anemia)
* Previous diagnosis not unequivocally resolved (chronic hepatitis, malignant tumors)
* Past neuropsychiatric disorders or current severe depressive disorder with psychotic or melancholy features, bipolar disorder, schizophrenia, delusional disorder, dementia, anorexia nervosa, bulimia nervosa
* Participation in another clinical trial of the same or different nature within 30 days prior to inclusion in the study
* Failure to provide signed informed consent
* Consumption of certain drugs/supplements that could affect outcome measures in the past 90 days or whose discontinuation could be a significant problem
* Anticoagulant treatment
* Pregnancy or breastfeeding
* Smoking, alcohol or substance abuse
* Obesity (BMI > 30 kg/m²)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
chronic fatigue symptoms | At baseline and after 3 months
  The primary outcome is the change in self-reported fatigue scores assessed using the Fatigue Impact Scale (FIS-40). The FIS-40 comprises 40 items divided into three domains (cognitive, physical, and psychosocial), each item scored from 0 (no fatigue) to 4 (severe fatigue). The total score ranges from 0 to 160, with higher scores indicating worse fatigue.

SECONDARY OUTCOMES:
Sleep quality | At baseline and after 3 months
  Sleep disturbances are assessed using the 19-item self-administered Pittsburgh Sleep Quality Index (PSQI) questionnaire. Scores are obtained on each of the seven sleep quality domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleeping pills, and daytime dysfunction. Each component is rated from 0 to 3 (0 = no sleep problems and 3 = severe sleep problems). The overall PSQI score ranges from 0 to 21 points, with scores ≥5 indicating worse sleep quality
Physical performance | At baseline and after 3 months
  Physical performance is assessed using the Short Physical Performance Battery test
Body composition | At baseline and after 3 months
  Body composition is assessed using the dual X-Ray absorptiometry (DXA)
Life quality | At baseline and after 3 months
  Quality of life is assessed using the Short-Form 12-Item Health Survey (SF-12), a short and generic measure of health status that reproduces the 2 summary scores of the SF-36. The summary of the physical component score and the summary score of the mental component, addressing eight health domains (physical functioning, physical role, body pain, general health, vitality, social functioning, emotional role, and mental health). Each domain is scored separately, and the total scores for the physical and mental components range from 0 to 100, with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- l'Istituto di Riabilitazione e cura "Santa Margherita" di Pavia, Azienda di Servizi alla Persona (ASP)., Pavia, Italy